CLINICAL TRIAL: NCT05320224
Title: Feasibility and Acceptability of a Patient-Oriented Music Intervention to Reduce Acute Pain in the Adult Intensive Care Unit: A Randomized Crossover Pilot Trial
Brief Title: Feasibility & Acceptability of a Patient-Oriented Music Intervention to Reduce Pain in the Intensive Care: A Pilot Trial
Acronym: POMI_PhaseII
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Céline Gélinas, Full Professor, Senior Researcher, McGill University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: POMI_Phase_II_2022_3005
Record Dates: First submitted 2022-03-10; First posted 2022-04-11 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Pain, Acute; Distress, Emotional; Critical Illness
MeSH Terms: conditions — Acute Pain; Critical Illness

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient-Oriented Music Intervention (POMI) followed by No Music - Sequence AB (Other): Patient participants will first receive 20-30 minutes of the patient-oriented music intervention (POMI) first, followed by no music, with a minimal washout period of four hours
  Interventions: Other: Patient-Oriented Music Intervention (POMI)
- No Music followed by Patient-Oriented Music Intervention (POMI) - Sequence BA (Other): Patient participants will first receive no music first, followed by 20-30 minutes of the patient-oriented music intervention (POMI), with a minimal washout period of four hours
  Interventions: Other: Patient-Oriented Music Intervention (POMI)

INTERVENTIONS:
Other: Patient-Oriented Music Intervention (POMI) — The brief name given to this intervention is POMI (Patient-Oriented Music Intervention). In POMI, music is delivered to adult patients either via headphones (Bose) or by music pillow (MusiCure). Adults admitted to the intensive care unit (ICU) will choose the mode of delivery. ICU adult patients who are unable to self-report will hear music via music pillow. Individualized playlists will be created based on the patient music preferences, as self-reported. For patients unable to self-report, a person significant to the patient such as a family member will be asked about the patient music preferences. Questions about preferences will include music genre, track, artist, instrumentalness, acousticness, energy, and valence, as defined by the streaming service Spotify. A POMI web-based tool (https://pomi.glitch.me) will use these preferences to create personalized playlists on Spotify, with a tempo restriction of 60-80 bpm. Music will play for at least 20 minutes, via smart device (iPad).

SUMMARY:
Introduction Many patients experience pain in the intensive care unit (ICU) despite receiving pain medication. Research has shown that music can help manage pain. Music interventions that have been studied so far have not been based on patient preferences, recommended tempo and duration, nor used music streaming. It is important that a music intervention take into consideration the expertise of ICU patients, family members and nurses/orderlies.

Study objectives This study aims to evaluate the feasibility and acceptability of a new patient-oriented music intervention (POMI) to reduce pain in ICU patients. In addition, the aim is to evaluate the feasibility of conducting a crossover randomized controlled trial (RCT) to test the interventions in the adult ICU. A secondary objective will be to examine the preliminary efficacy of the POMI.

Methodology/Study Design A single-blind 2x2 crossover pilot RCT will be used to evaluate the feasibility, acceptability, and preliminary efficacy of the POMI. Patients will undergo a sequence of two intervention periods: the POMI and the Active Control intervention (ACI; headphones/pillow without music). Patients will be randomly assigned to Sequence 1 or Sequence 2, where patients in Sequence 1 receive the POMI during the first intervention period, followed by the ACI in the second intervention period; and patients in Sequence 2 receive the ACI first, followed be the POMI (with a 4-hour washout period).

Before the turning procedure, music will be stopped, and the headphones will be removed. For patients able to self-report, the music (or control period without music) will be delivered either via headphones or a music pillow, depending on their individual preference. For patients unable to self-report, music (or control period without music) will be delivered via the music pillow.

Twenty-four patients (12 patients able to self-report their pain and 12 patients unable to self-report) will be recruited. The 12 patients able to self-report will be asked about their music preferences and to complete an acceptability questionnaire (AQ). For the 12 patients unable to self-report, 12 family members will be recruited to answer questions on the patient's music preferences and to complete an AQ. In addition, 12 nurses/orderlies (involved in the turning procedure for a patient participant) will be recruited and asked to complete an AQ.

ELIGIBILITY:
Inclusion criteria:

* ≥ 18 years old (all patients)
* Admitted to ICU (all patients)
* Able to self-report (patients able to self-report)
* Able to listen to music as per patient (patients able to self-report)
* Significant person is present at bedside (patients unable to self-report)
* Considers self to have knowledge of the patient's music preferences (significant persons)
* Is qualified to consent to any care required by the state of health for the incapable ICU adult patient (significant persons)
* Is present during turning procedure at the time of the POMI project data collection (nurses/orderlies)

Exclusion criteria:

* Cannot be turned (all patients)
* Does not speak/understand French or English (all participants)
* RASS -5 (all patients)
* Under effects of neuromuscular blocking agents (all patients)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-09-10 (Estimated); Study Completion 2022-09-10 (Estimated)

PRIMARY OUTCOMES:
Acceptability questionnaire, adapted from the validated Treatment Acceptability and Preferences questionnaire, 0-20 rating scores | 60 minutes
  The acceptability questionnaire is adapted from the validated Treatment Acceptability and Preferences (TAP) questionnaire. The TAP and is comprised of four items: suitability, appropriateness, effectiveness and willingness to comply, each of which is rated on a 5-point scale ranging from 0 (not at all) to 4 (very much) for a total score ranging from 0 to 20, with higher scores indicating higher acceptability. The total scale score is obtained by calculating the mean of all the items' scores. The TAP can capture the complex nature of participants' preferences and yet be simple enough for use in the ICU setting. One item has been added to the questionnaire to determine the risks of side effects of the POMI, an additional important aspect in assessing the acceptability of the intervention.
Feasibility of intervention delivery | up to 60 minutes
  The items for the assessment of the feasibility of intervention include time spent creating the individualized playlist, the presence or absence of any issue with headphone or pillow use, the presence or absence of any issue with music delivery, the presence or absence of skipping one or more song from the generated playlist, the presence or absence of any environmental noise, any POMI interruptions, whether the ICU adult patient participant received the full duration of the POMI, the dose (duration in minutes) of the music actually delivered, and the content of the music delivered (details of the music pieces played).

SECONDARY OUTCOMES:
Change from Baseline Pain intensity on the 11-point Numeric Rating Scale (NRS) at 30 minutes | Baseline and 30 minutes
  The Faces Pain Thermometer (FPT) is a 0-10 NRS with faces in a thermometer format allowing the measurement of self-reported pain intensity by patients. The FPT is advantageous for use in ICU adult patients not only for its concomitant use of faces with 0-10 number, but also for being presented vertically, facilitating the interpretation of the scale in adults of all ages. The FPT is reported to have acceptable test-retest reliability (Pearson's r, 0.63), high content validation (content validity indices, 0.73-1.00), high convergent validation with the descriptive pain scale (kappa coefficients ranging from 0.63-0.79) as well as discriminative validation, with significantly higher pain scores during nociceptive/painful events compared to non-nociceptive/non-painful events
Change from Baseline Pain intensity on the 11-point Numeric Rating Scale (NRS) at Bed Turning | From baseline to bed turning, up to 90 minutes
  The Faces Pain Thermometer (FPT) is a 0-10 NRS with faces in a thermometer format allowing the measurement of self-reported pain intensity by patients. The FPT is advantageous for use in ICU adult patients not only for its concomitant use of faces with 0-10 number, but also for being presented vertically, facilitating the interpretation of the scale in adults of all ages. The FPT is reported to have acceptable test-retest reliability (Pearson's r, 0.63), high content validation (content validity indices, 0.73-1.00), high convergent validation with the descriptive pain scale (kappa coefficients ranging from 0.63-0.79) as well as discriminative validation, with significantly higher pain scores during nociceptive/painful events compared to non-nociceptive/non-painful events
Change from Bed Turning Pain intensity on the 11-point Numeric Rating Scale (NRS) at 30 minutes | From bed turning (up to 90 minutes post baseline) to 30 minutes post bed turning
  The Faces Pain Thermometer (FPT) is a 0-10 NRS with faces in a thermometer format allowing the measurement of self-reported pain intensity by patients. The FPT is advantageous for use in ICU adult patients not only for its concomitant use of faces with 0-10 number, but also for being presented vertically, facilitating the interpretation of the scale in adults of all ages. The FPT is reported to have acceptable test-retest reliability (Pearson's r, 0.63), high content validation (content validity indices, 0.73-1.00), high convergent validation with the descriptive pain scale (kappa coefficients ranging from 0.63-0.79) as well as discriminative validation, with significantly higher pain scores during nociceptive/painful events compared to non-nociceptive/non-painful events
Change from Baseline Pain distress on the 11-point Numeric Rating Scale (NRS) at 30 minutes | Baseline and 30 minutes
  Evaluation of the affective dimension of pain will be conducted using the validated a 0-10 pain distress score, derived from the NRS, ranging from no distress (0) to very distressing (10). In a study conducted with 3851 patients across 28 countries across 192 adult ICUs, higher degrees of pain distress were associated with turning procedures (relative risk = 1.18) and turning procedures predicted greater pain distress than pain intensity (odds ratio = 0.626).
Change from Baseline Pain distress on the 11-point Numeric Rating Scale (NRS) at Bed Turning | From baseline to bed turning, up to 90 minutes
  Evaluation of the affective dimension of pain will be conducted using the validated a 0-10 pain distress score, derived from the NRS, ranging from no distress (0) to very distressing (10). In a study conducted with 3851 patients across 28 countries across 192 adult ICUs, higher degrees of pain distress were associated with turning procedures (relative risk = 1.18) and turning procedures predicted greater pain distress than pain intensity (odds ratio = 0.626).
Change from Bed Turning Pain distress on the 11-point Numeric Rating Scale (NRS) at 30 minutes | From bed turning (up to 90 minutes post baseline) to 30 minutes post bed turning
  Evaluation of the affective dimension of pain will be conducted using the validated a 0-10 pain distress score, derived from the NRS, ranging from no distress (0) to very distressing (10). In a study conducted with 3851 patients across 28 countries across 192 adult ICUs, higher degrees of pain distress were associated with turning procedures (relative risk = 1.18) and turning procedures predicted greater pain distress than pain intensity (odds ratio = 0.626).
Change from Baseline Critical-Care Pain Observation Tool (CPOT) at 30 minutes | Baseline and 30 minutes
  Evaluation of pain using the CPOT yields a score between zero and eight with scores above 2 representing the presence of pain. More specifically, the CPOT includes 4 items that can each be scored from 0-2: facial expression, body movements, muscle tension and vocalization/ventilator compliance. The CPOT has been validated in 47 studies with 3966 ICU patients unable to self-report across 21 different countries. Interrater reliability was examined in 30 studies, as determined by intra-class correlation and/or weighted kappa values above 0.60. Discriminative validation has been consistently supported with significantly higher CPOT scores during nociceptive/painful events compared to rest periods of rest or non-nociceptive/non-painful events, as evaluated by all studies that measured it (n = 43).
Change from Baseline Critical-Care Pain Observation Tool (CPOT) at Bed Turning | From baseline to bed turning, up to 90 minutes
  Evaluation of pain using the CPOT yields a score between zero and eight with scores above 2 representing the presence of pain. More specifically, the CPOT includes 4 items that can each be scored from 0-2: facial expression, body movements, muscle tension and vocalization/ventilator compliance. The CPOT has been validated in 47 studies with 3966 ICU patients unable to self-report across 21 different countries. Interrater reliability was examined in 30 studies, as determined by intra-class correlation and/or weighted kappa values above 0.60. Discriminative validation has been consistently supported with significantly higher CPOT scores during nociceptive/painful events compared to rest periods of rest or non-nociceptive/non-painful events, as evaluated by all studies that measured it (n = 43).
Change from Bed Turning Critical-Care Pain Observation Tool (CPOT) at 30 minutes | From bed turning (up to 90 minutes post baseline) to 30 minutes post bed turning
  Evaluation of pain using the CPOT yields a score between zero and eight with scores above 2 representing the presence of pain. More specifically, the CPOT includes 4 items that can each be scored from 0-2: facial expression, body movements, muscle tension and vocalization/ventilator compliance. The CPOT has been validated in 47 studies with 3966 ICU patients unable to self-report across 21 different countries. Interrater reliability was examined in 30 studies, as determined by intra-class correlation and/or weighted kappa values above 0.60. Discriminative validation has been consistently supported with significantly higher CPOT scores during nociceptive/painful events compared to rest periods of rest or non-nociceptive/non-painful events, as evaluated by all studies that measured it (n = 43).

CONTACTS AND LOCATIONS:
Overall Officials: Céline Gélinas, RN, PhD, Principal Investigator — McGill University
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Richard-Lalonde M, Feeley N, Cossette S, Chlan LL, Gelinas C. Acceptability and Feasibility of a Patient-Oriented Music Intervention to Reduce Pain in the Intensive Care Unit: Protocol for a Crossover Pilot Randomized Controlled Trial. JMIR Res Protoc. 2023 May 10;12:e40760. doi: 10.2196/40760. PMID 37163350